CLINICAL TRIAL: NCT06033469
Title: Therapeutic Monitoring of Infliximab and Adalimumab in Pediatric Chronic Inflammatory Diseases: Innovative Pharmacological Strategies for Predicting Response and Adverse Effects
Brief Title: Therapeutic Monitoring of Infliximab and Adalimumab
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 01/17
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Infliximab; Adalimumab; Inflammatory Bowel Diseases; Pharmacokinetics
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Infliximab; Adalimumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD group: Pediatric patients with IBD
  Interventions: Drug: Infliximab; Drug: Adalimumab

INTERVENTIONS:
Drug: Infliximab — Pediatric patients with IBD suitable for treatment with infliximab
Drug: Adalimumab — Pediatric patients with IBD suitable for treatment with adalimumab

SUMMARY:
Anti tumor necrosis factor (TNF agents), particularly infliximab and adalimumab, changed the way chronic inflammatory bowel disease (IBD) refractory to conventional therapies is treated, including in pediatric patients. However, approximately 10-30% of patients do not respond to initial therapy and up to 50% lose response over time. Variability in response to therapy may be influenced by multiple interacting factors at different levels. Recent studies showed that measurement of serum infliximab concentrations during induction therapy predicts treatment effects at one year. Therefore, therapeutic monitoring of infliximab is proposed as a useful strategy to improve clinical outcomes and optimize healthcare resources.

Most commercially available methods for infliximab quantification are based on the ELISA assay, which has an assay time of at least 8 hours. Recently, commercial point-of-care devices became available with assay times of less than one hour, enabling real-time therapeutic drug monitoring; however, validation of these devices in clinical settings and comparison with standard assays are still needed, particularly in pediatric patients. In addition, some studies suggest that loss of response in patients treated with anti-TNFs may be partly due to the emergence of specific anti-drug antibodies (AAFs). A limitation of the most widely used ELISA assays is the inability to quantify drug and AAF when they are simultaneously present. Recently, innovative ELISA assays have become available to overcome this problem. However, there is a lack of comparative studies between the classical and the specific method in terms of clinical response in pediatric patients. In patients who do not respond to infliximab, especially if they have high levels of AAF, guidelines call for the use of adalimumab. For this drug, the evidence in the literature regarding therapeutic monitoring of adalimumab concentrations and association with response in pediatric patients is still very preliminary. This study, carried out in in pediatric patients with IBD, aims to:

1. validate the "point of care" infliximab assay by comparing it with reference ELISA assays;
2. evaluate the correlation of infliximab and AAF levels, as measured by the innovative ELISA assays, with response to therapy, compared to traditional assays.
3. evaluate the association between adalimumab and AAF levels and response to therapy

DETAILED DESCRIPTION:
Anti-TNF agents, particularly infliximab and adalimumab, changed the way chronic inflammatory bowel disease (IBD) refractory to conventional therapies is treated, including in pediatric patients. These biologic agents also appear promising as first-line treatment even in the early stages of the disease. However, approximately 10-30% of patients do not respond to initial therapy and up to 50% lose response over time. In addition, the widespread use of these drugs is limited by serious side effects and the high cost of therapy. Variability in response to therapy may be influenced by multiple interacting factors at different levels. Recent studies showed that measurement of serum infliximab concentrations during induction therapy predicts treatment effects at one year: in particular, patients with infliximab concentrations below 3 ug/ml at the end of induction (pre-dose IV infusion) have a reduced probability of response. Therefore, therapeutic monitoring of infliximab is proposed as a useful strategy to improve clinical outcomes and optimize healthcare resources.

Currently, most commercially available methods for infliximab quantification are based on the ELISA assay, which has an assay time of at least 8 hours, delaying therapeutic adjustment to the next drug infusion. Recently, commercial point-of-care devices became available with assay times of less than one hour, enabling real-time therapeutic drug monitoring; however, validation of these devices in clinical settings and comparison with standard assays are still needed, particularly in pediatric patients. In addition, some studies suggest that loss of response in patients treated with anti-TNFs, infliximab and adalimumab, may be partly due to the emergence of specific anti-drug antibodies (AAFs). A limitation of the most widely used ELISA assays is the inability to quantify drug and AAF when they are simultaneously present. Data from the literature suggest that in patients who lose response to anti-TNFs, classical ELISA assays may overestimate the percentage of patients with low levels of both drug and AAF; the use of specific ELISA assays allows accurate quantification of drug and AAF levels even in these patients, allowing the clinician to modify therapy accordingly. Recently, innovative ELISA assays have become available to overcome this problem. However, there is a lack of comparative studies between the classical and the specific method in terms of clinical response in pediatric patients. In patients who do not respond to infliximab, especially if they have high levels of AAF, guidelines call for the use of adalimumab. For this drug, the evidence in the literature regarding therapeutic monitoring of adalimumab concentrations and association with response in pediatric patients is still very preliminary. Thus, the research objectives are three, of equal importance:

1. to validate the "point of care" infliximab assay by comparing it with reference ELISA assays in pediatric patients with IBD;
2. to evaluate the correlation of infliximab and AAF levels, as measured by the above innovative ELISA assays, with response to therapy, compared to traditional assays, in pediatric patients with IBD.
3. to evaluate the association between adalimumab and AAF levels and response to therapy in pediatric patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

* IBD subjects
* age between 0 and 17 years
* suitable for treatment with infliximab or adalimumab

Exclusion Criteria:

* Pediatric subjects with IBD not suitable for treatment with infliximab or adalimumab

Ages: 1 Year to 17 Years | Sex: All
Age Groups: Child
Study Population: Pediatric subjects with IBD suitable for treatment with infliximab or adalimumab
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Infliximab concentration | Through study completion, an average of 5 years
  Assessed with the point-of-care assay and with the ELISA assay
Adalimumab concentration | Through study completion, an average of 5 years
  Assessed with ELISA assay
AAF concentration | Through study completion, an average of 5 years
  Assessed by the novel ELISA assays
Response to therapy assessed with validated score | Through study completion, an average of 5 years
  Assessed by Pediatric Crohn's disease activity index (PCDAI) and Pediatric UlcerativeColitis Activity Index (PUCAI). PCDAI ranges from 0 to 100; higher scores indicate more active disease. Clinical remission was defined as PCDAI ≤ 10. PUCAI score ranges from 0 to 85, with disease remission less than 10, mild disease activity between 10-35, moderate disease activity from 35-65, and severe disease activity above 65

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Stocco, MSC, Principal Investigator — IRCCS materno infantile Burlo Garofolo
Locations (3):
- Italy (3):
  - Ospedale Maggiore, Bologna
  - Ospedale Ca' Foncello, Treviso
  - IRCCS Burlo Garofolo, Trieste